CLINICAL TRIAL: NCT06542861
Title: Effects of in Situ Simulation-based Team Training on Clinical Performance During Pediatric Cardiac Arrest: An Intervention Study Comparing Two Danish Regions
Brief Title: Effects of High-Frequency In Situ Simulation-based Team Training on Clinical Performance During Pediatric Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Corporate HR, MidtSim, Central Denmark Region (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1-16-02-77-23
Record Dates: First submitted 2024-06-19; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-04

CONDITIONS: Medical Education; Simulation-based Training; In-hospital Cardiac Arrest; Pediatrics; in Situ Simulation
Keywords: In-hospital cardiac arrest; Medical Education; Simulation-based training; Pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Healthcare professionals (doctors and nurses) employed in one of four pediatric departments in the Central Denmark Region. N = approximately 600.
  From April 1st 2023 to April 1st 2024 healthcare professionals in the intervention arm will be exposed to a high-frequency training program, in which each healthcare professional will attend four SBTT sessions in one year, approx. three months apart. Three-month intervals were chosen based on knowledge of retention of technical skills.
  Interventions: Other: High-frequency simulation-based team training
- Control (No Intervention): Healthcare professionals (doctors and nurses) employed in one of four pediatric departments in the Region of Southern Denmark. N = approximately 600.
  No special training program. Participants in the control region will continue simulation-based team training "as usual" with no changes in training frequency.

INTERVENTIONS:
Other: High-frequency simulation-based team training — The intervention is a standardized high-frequency training program as described in intervention arm. It is supported by four preliminary initiatives:
  1. 15 extra pediatric simulation facilitators were educated, bringing the total number up to 40.
  2. A two-day pre-intervention workshop for all pediatric simulation facilitators.
  3. A "scenario bank" containing standardized scenarios on common pediatric and neonatal emergencies was created and made accessible for simulation facilitators to support consistency in the intervention.
  4. Purchase of equipment. Eight Leardal manikins. Four SimPads. Four monitors. During the intervention year, these will rotate between the pediatric departments.
  Arms: Intervention

SUMMARY:
Cardiac arrest in hospitalized children is a rare occurrence in general and for each healthcare professional in particular, making lack of routine in performing cardiopulmonary resuscitation a challenge. Mortality and morbidity following cardiac arrest depend on the technical (medical knowledge, procedures, etc.) and non-technical (team leadership, communication, etc.) skills performed by the medical team. Simulation-based team training is a well-known and effective method to improve team performance in high-stake and time-sensitive situations, without putting actual patients at risk. Unfortunately, studies show that skills obtained during simulation-based team training decline within a few months. However, recent observational studies have demonstrated improved technical pediatric basic life support skills after short simulation sessions with a high frequency of repeat. The healthcare professionals in these studies are limited to selected groups and tests are performed exclusively on skill stations.

In this study, the effects of a novel high-frequency training program will be investigated. A controlled intervention study in two comparable Danish regions will be conducted. Healthcare professionals in four pediatric departments in the intervention region will participate in the high-frequency training program. Healthcare professionals in four pediatric departments in the control region will continue simulation-based team training with no changes - "as usual" and at a two to three times lower frequency (based on unpublished data). Both groups consist of approximately 600 healthcare professionals, contributing to a total of 1,200 participants included in this project.

Hypotheses: high-frequency training will improve primary outcomes during in-situ simulated pediatric in-hospital cardiac arrest as specified:

1. Teamwork competencies measured by the team emergency assessment measure (TEAM),
2. Time (seconds) to recognition of cardiac arrest.
3. Time (seconds) to initiation of cardiopulmonary resuscitation.
4. Longest chest compression pause duration.

Data collection. To assess clinical performance in both regions unannounced in-situ (in own department with usage of own equipment) simulations of pediatric cardiac arrest will be performed and recorded on video.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (doctor or nurse) employed in one of the eight pediatric departments in Central Denmark Region og Southern Denmark Region during the project period April 1st 2023 to April 1st 2024.

Exclusion Criteria:

* Missing consent to be recorded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Teamwork competences | Up to 36 months
  Global team score. Assessed in both regions pre- and post-intervention. Assessed according to Team Emergency Assessment Measure (TEAM). Score range from 1-54. 1 being the lowest score and 54 the highest.
Time to diagnosis of cardiac arrest | Up to 36 months
  Time (seconds) until cardiac arrest is recognized, assessed in both regions by pre- and post-intervention video recordings of unannounced in-situ simulations of pediatric cardiac arrest.
Time to initiation of cardiopulmonary resuscitation | Up to 36 months
  Time (seconds) until cardiopulmonary resuscitation within standard guidelines for neonates/children is initiated, assessed in both regions by pre- and post-intervention video recordings of unannounced in-situ simulations of pediatric cardiac arrest.
Longest chest compression pause duration | Up to 36 months
  Chest compression pause durations will be assessed in both regions by pre- and post-intervention video recordings of unannounced in-situ simulations of pediatric cardiac arrest.

SECONDARY OUTCOMES:
Team effectiveness | Up to 36 months.
  Time (seconds) to: call for help, arrival of defibrillator, first rhythm check. Will be assessed in both regions by pre- and post-intervention video recordings of unannounced in-situ simulations of pediatric cardiac arrest.
Cardiopulmonary resuscitation quality | Up to 36 months.
  Proportion of compressions, and ventilations within guideline recommendations for depth/rate and tidal volumes, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Morten S Lindhard, MD, PhD, Study Director — Randers Regional Hospital
Locations (1):
- Corporate HR, MidtSim, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT06542861/Prot_000.pdf